CLINICAL TRIAL: NCT00983060
Title: A Randomized, Adaptive-design, Dose-finding Study to Assess the Antiviral Efficacy and Safety of NIM811 Administered in Combination With the Standard of Care (SOC) in Relapsed Patients Infected With HCV Genotype-1
Brief Title: Adaptive-design Dose Finding Study to Assess the Antiviral Efficacy and Safety of NIM811 Administered in Combination With Standard of Care (SOC) in Relapsed Hepatitis C Virus 1 (HCV-1) Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNIM811B2202; EUDRACT number: 2009-009995-11
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-02

CONDITIONS: Chronic Hepatitis C Genotype-1 Relapse
Keywords: NIM811; chronic hepatitis; chronic hepatitis C; chronic hepatitis C genotype-1; HCV; HCV-1; relapser
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis C, Chronic | interventions — (melle-4)cyclosporin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- NIM811 (Experimental)
  Interventions: Drug: NIM811
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo BID + SOC

INTERVENTIONS:
Drug: NIM811 — BID in various doses (between 100 mg - 600 mg bid) + SOC (PEG IFN and RBV)
  Arms: NIM811
Drug: Placebo BID + SOC — Placebo BID + SOC (PEG IFN and RBV)
  Arms: Placebo

SUMMARY:
This is a study designed to identify a dose of NIM811 that has a good safety profile, is well tolerated when co-administered with SOC, and provides a clinically meaningful effect in viral load reduction compared to SOC alone. This information will be used to support doses selected for future studies.

ELIGIBILITY:
Inclusion criteria:

Patients eligible for inclusion in this study have to fulfill all of the following criteria:

* chronic hepatitis C genotype-1
* HCV-RNA should be ≥ 4 x 105 IU/mL at screening
* Recipient of prior long acting interferon and ribavirin treatment for at least 12 weeks, with documented negative serum HCV RNA on treatment, who subsequently becomes serum HCV RNA positive after stopping treatment ("relapser"). Patients must have been off all treatment for at least 3 months prior to start of study (Visit

Exclusion criteria:

* Use of any HCV treatment ≤ 3months prior to study start
* Prior receipt of any investigational anti-HCV therapy which is not IFN or RBV
* Women of child-bearing potential unless they are post-menopausal or use predefined acceptable methods of contraception
* Pregnant or breastfeeding women
* Evidence of cirrhosis, hepatic decompensation, other than HCV liver disease, HBV or HIV infection
* Specified abnormalities in lab values of amongst others hemoglobin, WBC, ANC, platelets
* History of treatment for depression
* Steroid/immunosuppression drug use 3 months prior to study start Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of NIM811 dosed daily for 4 weeks in combination with SOC | 4 weeks

SECONDARY OUTCOMES:
To identify a dose of NIM811 which is safe and tolerated and produces in combination with SOC a clinically meaningful improvement over SOC monotherapy in antiviral response Time Frame: 4 weeks | 12 weeks
To assess the percentage of patients achieving rapid virologic response (RVR) in patients treated with NIM811 in combination with SOC | 4 weeks
To explore the pharmacokinetics and pharmacodynamics of NIM811 given in combination with SOC in patients with chronic hepatitis C genotype-1 | 3 weeks, 5 weeks
To evaluate the effect of NIM811 given in combination with SOC in patients with chronic hepatitis C genotype-1 on sustained virologic response 12 weeks after cessation of treatment (SVR12) | 12 weeks after cessation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (5):
  - Research and Education Inc., San Diego, California
  - Orlando Clinical Research Center, Orlando, Florida
  - University Hepatitis Center, Sarasota, Florida
  - West Wind'r Research & Development LLC, Tampa, Florida
  - Alamo Medical Research, San Antonio, Texas
- Australia (3):
  - Novartis Investigative Site, Clayton, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Wentworthville, South Australia
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Frankfurt, Germany
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Seville
- Taiwan (2):
  - Novartis Investigative Site, Taipei, ROC
  - Novartis Investigative Site, Kaohsiung City

REFERENCES:
- [Result] Lawitz E, Godofsky E, Rouzier R, Marbury T, Nguyen T, Ke J, Huang M, Praestgaard J, Serra D, Evans TG. Safety, pharmacokinetics, and antiviral activity of the cyclophilin inhibitor NIM811 alone or in combination with pegylated interferon in HCV-infected patients receiving 14 days of therapy. Antiviral Res. 2011 Mar;89(3):238-45. doi: 10.1016/j.antiviral.2011.01.003. Epub 2011 Jan 19. PMID 21255610
- See also: Results for CNIM811B2202 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6083